CLINICAL TRIAL: NCT00404469
Title: Effects of Peritendinous Corticosteroid Injections, Eccentric Training and Heavy Slow Resistance Training in Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Patellar tendinopathy
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Patellar Tendinopathy / Jumpers Knee

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- CORT (Active Comparator): Peritendinous corticosteroid injections at 0 and 4 weeks. 12 weeks total
  Interventions: Procedure: peritendinous corticosteroid injections
- ECC (Experimental): 12 weeks of eccentric unilateral decline squats
  Interventions: Procedure: eccentric decline squat training
- HSR (Experimental): Heavy slow resistance training. 3/week. 12 weeks
  Interventions: Procedure: heavy slow resistance training

INTERVENTIONS:
Procedure: peritendinous corticosteroid injections — 1 ml of40mg/ml methylprednisolone acetate at 0 and 4 weeks. 2 week observational
  Arms: CORT
Procedure: eccentric decline squat training — eccentric decline unilateral squats performed twice daily. for 12 weeks
  Arms: ECC
Procedure: heavy slow resistance training — Heavy slow resistance training for knee extensors. 3/week. total of 12 weeks
  Arms: HSR

SUMMARY:
We will investigate the effect of peritendinous corticosteroid injections, eccentric training and heavy resistance training in male patellar tendinopathy patients. The purpose is to compare the clinical effect of these three treatments in a randomised controlled trial. Also we wish to investigate the treatment mechanisms responsible for the effectiveness of the three treatments.

DETAILED DESCRIPTION:
3 interventions groups as described above (n=13 in each group) 12 weeks intervention period. Clinical assessments before and after intervention: VAS, VISA, Tendon thickness, Doppler us activity.

Before and after intervention tendon biopsies will be taken and analyzed for crosslinks and fibril diameter. Also tendon mechanical properties will be measured. Tendon and muscle structural properties will be measured with MRI.

Treatment satisfaction will be stated after intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical patellar tendinopathy pain.
* Tendon swelling
* Hypoechoic
* Doppler activity in tendon

Exclusion Criteria:

* Previous knee surgery
* diabetes
* arthritis
* previous steroid injections

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-03; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mads Kongsgaard, PhD., MSc., Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen. Dept 8 1st floor. Bispebjerg Hospital, Copenhagen, Denmark